CLINICAL TRIAL: NCT05869734
Title: Effects of Conservative Management Incorporating Urologic Health Promotion and Sleep Health Promotion on Relieving Storage Urinary Symptoms and Poor Sleep in Women With Diabetes
Brief Title: Effects of Conservative Management on Relieving Storage Urinary Symptoms and Poor Sleep in Women With Diabetes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Collaborators: Cardinal Tien Hospital (Other)
Responsible Party: Principal Investigator, Yuan-Mei Liao, RN, PhD, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11131006
Record Dates: First submitted 2023-04-26; First posted 2023-05-22 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Conservative Management; Diabetes Mellitus; Health-related Quality of Life; Lower Urinary Tract Symptoms; Self-management; Sleep; Sleep Health
MeSH Terms: conditions — Diabetes Mellitus; Lower Urinary Tract Symptoms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group A (Experimental): The intervention group A receives conservative management with sleep hygiene related adjustments, pelvic floor muscle training, and urologic health promotion.
  Interventions: Behavioral: Sleep health promotion; Behavioral: Urologic health promotion; Behavioral: Pelvic floor muscle training
- Intervention group B (Experimental): The intervention group B receives conservative management with brief behavioral treatment for insomnia (BBTI), pelvic floor muscle training, and urologic health promotion.
  Interventions: Behavioral: Sleep health promotion; Behavioral: Urologic health promotion; Behavioral: Pelvic floor muscle training
- Comparison group (Sham Comparator): The comparison group receives information related to pelvic floor muscle training and urologic health promotion.
  Interventions: Behavioral: Urologic health promotion; Behavioral: Pelvic floor muscle training

INTERVENTIONS:
Behavioral: Sleep health promotion — We will provide sleep hygiene related adjustments in the intervention group A; and brief behavioral treatment for insomnia (BBTI) in the intervention group B.
  Arms: Intervention group A; Intervention group B
Behavioral: Urologic health promotion — We will provide information related to urologic health promotion in three groups (2 experimental groups and 1 comparison group).
Behavioral: Pelvic floor muscle training — We will provide information related to pelvic floor muscle training in three groups (2 experimental groups and 1 comparison group).

SUMMARY:
Women with type 2 diabetes (n=90) experiencing ≥1 storage lower urinary tract symptoms and poor sleep health will be recruited from the outpatient departments or wards/units of the selected hospitals/clinics. Our study aims to examine the effects of conservative management incorporating urologic health promotion and sleep health promotion on relieving storage lower urinary tract symptoms and poor sleep, and on improving urologic health self-management behaviors and health-related quality of life. Women who agree to participate will be randomly assigned into the intervention group A, intervention group B, or comparison group. The intervention group A receives a 4-month conservative management with sleep hygiene related adjustments, pelvic floor muscle training, and urologic health promotion. The intervention group B receives a 4-month conservative management with brief behavioral treatment for insomnia (BBTI), pelvic floor muscle training, and urologic health promotion. The comparison group receives information related to pelvic floor muscle training and urologic health promotion, and receives a brief conservative management related to sleep hygiene adjustments after the completion of data collection. Information related to intervention effects is obtained by a questionnaire, a wristwatch-like actigraphy, and physical activity/diet/voiding/sleep logs from all participants at 4 data collection points: baseline, and 2-, 4-, 6-month follow-ups. Our study hypothesis is that the intervention effects on relieving storage lower urinary tract symptoms and poor sleep, and on improving urologic health self-management behaviors and health-related quality of life in the intervention group A or B are superior to the changes revealed in the comparison group.

DETAILED DESCRIPTION:
Women with type 2 diabetes (n=90) experiencing ≥1 storage lower urinary tract symptoms and poor sleep health will be recruited from the outpatient departments or wards/units of the selected hospitals/clinics. Our study aims to examine the effects of conservative management incorporating urologic health promotion and sleep health promotion on relieving storage lower urinary tract symptoms and poor sleep, and on improving urologic health self-management behaviors and health-related quality of life. Women who agree to participate will be randomly assigned into the intervention group A, intervention group B, or comparison group. The intervention group A receives a 4-month conservative management with sleep hygiene related adjustments, pelvic floor muscle training, and urologic health promotion. The intervention group B receives a 4-month conservative management with brief behavioral treatment for insomnia (BBTI), pelvic floor muscle training, and urologic health promotion. The comparison group receives information related to pelvic floor muscle training and urologic health promotion, and receives a brief conservative management related to sleep hygiene adjustments after the completion of data collection. Information related to intervention effects is obtained by a questionnaire, a wristwatch-like actigraphy, and physical activity/diet/voiding/sleep logs from all participants at 4 data collection points: baseline, and 2-, 4-, 6-month follow-ups. Our study hypothesis is that the intervention effects on relieving storage lower urinary tract symptoms and poor sleep, and on improving urologic health self-management behaviors and health-related quality of life in the intervention group A or B are superior to the changes revealed in the comparison group. The effects of the provided intervention on storage lower urinary tract symptoms, sleep quality, urologic health self-management behaviors, and health-related quality of life will be examined by Generalized Estimating Equations procedures with the estimations of effect sizes. Results of Chi-squared tests and descriptive statistics will also be used to present the intervention effects.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age 50-79 years
* Clinical diagnosis of diabetes >3 months
* Experiencing ≥1 storage lower urinary tract symptoms in the past 1 month
* Experiencing poor sleep health in the past 1 month
* Intact cognition and communication abilities

Exclusion Criteria:

* Receiving urologic problems related treatments in the past 3 months
* Receiving sleep problems related treatments in the past 3 months
* Receiving mental problems related treatments in the past 3 months
* Having a history of spinal surgery, cardiovascular, renal, or nervous system diseases
* Having severe mental illness
* Having physical impairments

Ages: 20 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Lower urinary tract symptoms | Baseline
  We will use a lower urinary tract symptoms scale to assess eight common female lower urinary tract symptoms: nocturia, urinary incontinence, increased daytime urinary frequency, urgency, a slow stream, an intermittent stream, hesitancy, and a feeling of incomplete emptying. The total lower urinary tract symptoms score ranges from 0 to 8; a higher total score indicates an individual experiencing more types of lower urinary tract symptoms.
Lower urinary tract symptoms | The 2-month follow-up.
  We will use a lower urinary tract symptoms scale to assess eight common female lower urinary tract symptoms: nocturia, urinary incontinence, increased daytime urinary frequency, urgency, a slow stream, an intermittent stream, hesitancy, and a feeling of incomplete emptying. The total lower urinary tract symptoms score ranges from 0 to 8; a higher total score indicates an individual experiencing more types of lower urinary tract symptoms.
Lower urinary tract symptoms | The 4-month follow-up.
  We will use a lower urinary tract symptoms scale to assess eight common female lower urinary tract symptoms: nocturia, urinary incontinence, increased daytime urinary frequency, urgency, a slow stream, an intermittent stream, hesitancy, and a feeling of incomplete emptying. The total lower urinary tract symptoms score ranges from 0 to 8; a higher total score indicates an individual experiencing more types of lower urinary tract symptoms.
Lower urinary tract symptoms | The 6-month follow-up.
  We will use a lower urinary tract symptoms scale to assess eight common female lower urinary tract symptoms: nocturia, urinary incontinence, increased daytime urinary frequency, urgency, a slow stream, an intermittent stream, hesitancy, and a feeling of incomplete emptying. The total lower urinary tract symptoms score ranges from 0 to 8; a higher total score indicates an individual experiencing more types of lower urinary tract symptoms.
Sleep Quality | Baseline.
  Sleep quality will be measured by the Chinese version of the Pittsburgh Sleep Quality Index. The Chinese version of the Pittsburgh Sleep Quality Index score ranges from 0 to 21; a lower Chinese version of the Pittsburgh Sleep Quality Index score indicates an individual experiencing better subjective sleep quality.
Sleep Quality | The 2-month follow-up.
  Sleep quality will be measured by the Chinese version of the Pittsburgh Sleep Quality Index. The Chinese version of the Pittsburgh Sleep Quality Index score ranges from 0 to 21; a lower Chinese version of the Pittsburgh Sleep Quality Index score indicates an individual experiencing better subjective sleep quality.
Sleep Quality | The 4-month follow-up.
  Sleep quality will be measured by the Chinese version of the Pittsburgh Sleep Quality Index. The Chinese version of the Pittsburgh Sleep Quality Index score ranges from 0 to 21; a lower Chinese version of the Pittsburgh Sleep Quality Index score indicates an individual experiencing better subjective sleep quality.
Sleep Quality | The 6-month follow-up.
  Sleep quality will be measured by the Chinese version of the Pittsburgh Sleep Quality Index. The Chinese version of the Pittsburgh Sleep Quality Index score ranges from 0 to 21; a lower Chinese version of the Pittsburgh Sleep Quality Index score indicates an individual experiencing better subjective sleep quality.
Total nighttime sleep | Baseline.
  Total nighttime sleep will be measured by a wristwatch-like actigraphy. A longer total nighttime sleep duration indicates an individual having better sleep.
Total nighttime sleep | The 2-month follow-up.
  Total nighttime sleep will be measured by a wristwatch-like actigraphy. A longer total nighttime sleep duration indicates an individual having better sleep.
Total nighttime sleep | The 4-month follow-up.
  Total nighttime sleep will be measured by a wristwatch-like actigraphy. A longer total nighttime sleep duration indicates an individual having better sleep.
Total nighttime sleep | The 6-month follow-up.
  Total nighttime sleep will be measured by a wristwatch-like actigraphy. A longer total nighttime sleep duration indicates an individual having better sleep.
Sleep onset latency | Baseline.
  Sleep onset latency, the length of time that it takes to fall asleep, will be measured by a wristwatch-like actigraphy. A shorter sleep onset latency indicates that an individual is easier to fall asleep.
Sleep onset latency | The 2-month follow-up.
  Sleep onset latency, the length of time that it takes to fall asleep, will be measured by a wristwatch-like actigraphy. A shorter sleep onset latency indicates that an individual is easier to fall asleep.
Sleep onset latency | The 4-month follow-up.
  Sleep onset latency, the length of time that it takes to fall asleep, will be measured by a wristwatch-like actigraphy. A shorter sleep onset latency indicates that an individual is easier to fall asleep.
Sleep onset latency | The 6-month follow-up.
  Sleep onset latency, the length of time that it takes to fall asleep, will be measured by a wristwatch-like actigraphy. A shorter sleep onset latency indicates that an individual is easier to fall asleep.
Wake after sleep onset | Baseline.
  Wake after sleep onset, the amount of time scored as wake between sleep onset and sleep offset, will be measured by a wristwatch-like actigraphy. A shorter wake after sleep onset indicates an individual having better sleep.
Wake after sleep onset | The 2-month follow-up.
  Wake after sleep onset, the amount of time scored as wake between sleep onset and sleep offset, will be measured by a wristwatch-like actigraphy. A shorter wake after sleep onset indicates an individual having better sleep.
Wake after sleep onset | The 4-month follow-up.
  Wake after sleep onset, the amount of time scored as wake between sleep onset and sleep offset, will be measured by a wristwatch-like actigraphy. A shorter wake after sleep onset indicates an individual having better sleep.
Wake after sleep onset | The 6-month follow-up.
  Wake after sleep onset, the amount of time scored as wake between sleep onset and sleep offset, will be measured by a wristwatch-like actigraphy. A shorter wake after sleep onset indicates an individual having better sleep.
Sleep efficiency | Baseline.
  Sleep efficiency will be measured by a wristwatch-like actigraphy. Sleep efficiency is calculated as the ratio of total nighttime sleep to total time in bed multiplied by 100. A higher sleep efficiency (0 to 100) indicates an individual having better objective sleep quality.
Sleep efficiency | The 2-month follow-up.
  Sleep efficiency will be measured by a wristwatch-like actigraphy. Sleep efficiency is calculated as the ratio of total nighttime sleep to total time in bed multiplied by 100. A higher sleep efficiency (0 to 100) indicates an individual having better objective sleep quality.
Sleep efficiency | The 4-month follow-up.
  Sleep efficiency will be measured by a wristwatch-like actigraphy. Sleep efficiency is calculated as the ratio of total nighttime sleep to total time in bed multiplied by 100. A higher sleep efficiency (0 to 100) indicates an individual having better objective sleep quality.
Sleep efficiency | The 6-month follow-up.
  Sleep efficiency will be measured by a wristwatch-like actigraphy. Sleep efficiency is calculated as the ratio of total nighttime sleep to total time in bed multiplied by 100. A higher sleep efficiency (0 to 100) indicates an individual having better objective sleep quality.

SECONDARY OUTCOMES:
Health-related quality of life | Baseline.
  The Short Form-36 Health Survey including a probe of self-perceived changes in health (1 item) and 35 items belonged to eight aspects will be used to measure health-related quality of life. The eight aspect scores (0 to100) will be used to calculate the physical and mental component summary scores. A higher aspect score indicates an individual having a better health-related quality of life on that aspect; a higher physical or mental component summary score indicates an individual having a superior combination of physical or mental functions.
Health-related quality of life | The 2-month follow-up.
  The Short Form-36 Health Survey including a probe of self-perceived changes in health (1 item) and 35 items belonged to eight aspects will be used to measure health-related quality of life. The eight aspect scores (0 to100) will be used to calculate the physical and mental component summary scores. A higher aspect score indicates an individual having a better health-related quality of life on that aspect; a higher physical or mental component summary score indicates an individual having a superior combination of physical or mental functions.
Health-related quality of life | The 4-month follow-up.
  The Short Form-36 Health Survey including a probe of self-perceived changes in health (1 item) and 35 items belonged to eight aspects will be used to measure health-related quality of life. The eight aspect scores (0 to100) will be used to calculate the physical and mental component summary scores. A higher aspect score indicates an individual having a better health-related quality of life on that aspect; a higher physical or mental component summary score indicates an individual having a superior combination of physical or mental functions.
Health-related quality of life | The 6-month follow-up.
  The Short Form-36 Health Survey including a probe of self-perceived changes in health (1 item) and 35 items belonged to eight aspects will be used to measure health-related quality of life. The eight aspect scores (0 to100) will be used to calculate the physical and mental component summary scores. A higher aspect score indicates an individual having a better health-related quality of life on that aspect; a higher physical or mental component summary score indicates an individual having a superior combination of physical or mental functions.
Self-management of urologic health | Baseline.
  The self-management of urologic health scale will be used to measure self-management behaviors relating to urologic health promotion. A higher scale score indicates an individual having better urologic health self-management behaviors.
Self-management of urologic health | The 2-month follow-up.
  The self-management of urologic health scale will be used to measure self-management behaviors relating to urologic health promotion. A higher scale score indicates an individual having better urologic health self-management behaviors.
Self-management of urologic health | The 4-month follow-up.
  The self-management of urologic health scale will be used to measure self-management behaviors relating to urologic health promotion. A higher scale score indicates an individual having better urologic health self-management behaviors.
Self-management of urologic health | The 6-month follow-up.
  The self-management of urologic health scale will be used to measure self-management behaviors relating to urologic health promotion. A higher scale score indicates an individual having better urologic health self-management behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Yuan-Mei Liao, PhD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- Cardinal Tien Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No